CLINICAL TRIAL: NCT02733419
Title: Open-label, Randomised and Multi-center Study Evaluating the Efficacy and Safety of an Optimised Background Antiretroviral Regimen (OB) Compared to OB Associated With Enfuvirtide in Previously Treated HIV-1 Infected Patients in Virological Success After a 28-week Induction Treatment With Enfuvirtide Plus OB
Brief Title: Efficacy, and Safety Study of Optimized Background Antiretroviral Regimen (OB) in Combination With Enfuvirtide in the Treatment-Experienced Participants With Human Immunodeficiency Virus-1 (HIV-1) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18242
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (3):
- Enfuvirtide + OB (Not Randomized) (Experimental): Participants will receive enfuvirtide 90 milligram (mg) twice daily (b.i.d.) and OB as per investigator's discretion for 28 weeks during induction period. After induction period participants not meeting the randomization criteria will receive enfuvirtide 90 mg b.i.d and OB for next 24 weeks (up to Week 52).
  Interventions: Drug: Enfuvirtide; Drug: Optimized background antiretroviral regimen (OB)
- Enfuvirtide + OB (Randomized) (Experimental): Participants will receive enfuvirtide 90 mg b.i.d. and OB as per investigator's discretion for 28 weeks during induction period. After induction period participants meeting the randomization criteria will be randomized to receive enfuvirtide 90 mg b.i.d. and OB for next 24 weeks (up to Week 52).
  Interventions: Drug: Enfuvirtide; Drug: Optimized background antiretroviral regimen (OB)
- OB alone (Randomized) (Experimental): Participants will receive enfuvirtide 90 mg b.i.d. and OB as per investigator's discretion for 28 weeks during induction period. After induction period participants meeting the randomization criteria will be randomized to receive OB alone for next 24 weeks (up to Week 52).
  Interventions: Drug: Enfuvirtide; Drug: Optimized background antiretroviral regimen (OB)

INTERVENTIONS:
Drug: Enfuvirtide — Participants will receive 90 mg enfuvirtide subcutaneously (SC) b.i.d.
  Other Names: Fuzeon
Drug: Optimized background antiretroviral regimen (OB) — Participants will receive OB (nucleoside and or non-nucleoside reverse transcriptase inhibitor and protease inhibitor) as per investigator's discretion. Protocol does not specify any particular OB drugs.

SUMMARY:
This is an open-label, randomized and multi-center study to compare the efficacy and safety of continued enfuvirtide (Fuzeon) plus (+) OB therapy versus OB alone in participants with HIV-1 infection. Participants will receive an initial 28 week induction treatment with enfuvirtide + OB. After 28 weeks participants with a plasma viral load less than or equal to (</=) 400 copies/milliliter (mL) at Week 16 and less than (<) 50 copies/mL at Week 24 will be randomized in the ratio 1:1 to receive either enfuvirtide + OB or OB alone for another 24 weeks (up to Week 52).

ELIGIBILITY:
Inclusion Criteria:

* Participants with HIV-1 infection
* Female participants without any risk of pregnancy
* Participants previously treated with drugs of 2 or 3 different antiretroviral classes
* Participants currently on highly active antiretroviral treatment (HAART) for more than 4 weeks and with a plasma viral load between 1,000 and 300,000 copies of HIV-1 ribonucleic acid per milliliter (RNA/mL)
* Participants with the possibility of potentially effective OB without enfuvirtide, consisting to 2 to 5 drugs, at least two of which are active from at least two different antiretroviral classes
* Cluster of differentiation 4 (CD4) cell count greater than (>) 50 cells/cubic millimeter (mm^3) at screening
* Participants in whom resistance mutations have been detected in reverse transcriptase and/or protease genes
* Enfuvirtide-naive participants

Exclusion Criteria:

* Women of childbearing age not using effective mechanical contraception
* Pregnant or breastfeeding women
* Presence of HIV-2 coinfection
* Participants participating or having participated to another clinical trial during the 30 days prior to selection for this trial
* Participants having previously been treated with enfuvirtide
* Presence active opportunistic infection within 1 month of study entry
* Existence of Grade 4 clinical or laboratory abnormalities
* Cirrhosis or severe hepatic failure
* Uncontrolled diabetes or requiring insulin
* Consumption of alcohol and/or narcotics and/or other substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Percentage of randomized participants without virologic failure and with a viral load < 50 copies/mL at Week 52 | Week 52

SECONDARY OUTCOMES:
Number of participants with virologic response (viral load < 50 copies/mL, 200 copies/mL, and 400 copies/mL) | Weeks 2, 4, 8, 12, 16, 24, 28, 32, 36, 44, and 52
Number of participants who complied with enfuvirtide and OB treatments as measured by pharmacokinetic score | Weeks 2, 4, 8, and 24
Quality of life as assessed by medical outcomes study-HIV (MOS-HIV) questionnaire score | Day 0 (inclusion), Weeks 4, 12, 24, 28, 32, 44, and 52 or premature withdrawal
Change from baseline in viral load | Baseline up to Week 52 or premature withdrawal
Proviral deoxyribonucleic acid (DNA) level | Day 0 (inclusion), Weeks 28, and 52 or premature withdrawal
Time to reappearance of viral load above 50 copies/mL in randomized participants | 52 weeks
Changes from baseline in CD4 and CD8 cell counts | Day -35 (screening), Day 0 (inclusion), Weeks 4, 12, 24, 28, 36, 44, and 52 or premature withdrawal
Number of virologic failure participants with reverse transcriptase, protease, and coating resistance mutations for plasma HIV-1 RNA and proviral DNA | Day 0 (inclusion) up to Week 52
Number of participants with cause of virologic failure | Day 0 (inclusion), Weeks 2, 4, 8, 16, 28, 32, 36, 44, and 52 or premature withdrawal
Number of participants who complied with enfuvirtide treatment, as assessed by counting treatment units returned versus supplied | Weeks 4, 8, 12, 16, 24, 28, 32, 36, 44, and 52
Number of participants with adverse events | Day 0 (inclusion), Weeks 2, 4, 8, 12, 16, 24, 28, 32, 36, 44, and 52 or premature withdrawal and follow-up (approximately up to 452 days)
Number of participants with missed treatment doses or injections as assessed by compliance questionnaire | Day 0 (inclusion), Weeks 4, 12, 24, 28, 32, 44, and 52 or premature withdrawal
Number of participants with injection site reaction | Day 0 (inclusion), Weeks 2, 4, 8, 12, 16, 24, 28, 32, 36, 44, and 52 or premature withdrawal and follow-up (approximately up to 452 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (56):
- France (56):
  - Aix-en-Provence
  - Angers
  - Annecy
  - Argenteuil
  - Auch
  - Aulnay-sous-Bois
  - Avignon
  - Basse-terre
  - Besançon
  - Bobigny
  - Bordeaux
  - Boulogne
  - Bourg-en-Bresse
  - Caen
  - Carpentras
  - Cayenne
  - Colmar
  - Corbeil-Essonnes
  - Créteil
  - Fort-de-france
  - Garches
  - Kourou
  - La Roche-sur-Yon
  - Lagny-sur-Marne
  - Levallois-Perret
  - Lyon
  - Mantes-la-Jolie
  - Marseille
  - Matoury
  - Mâcon
  - Montpellier
  - Nantes
  - Nice
  - Niort
  - Nîmes
  - Orléans
  - Paris
  - Pau
  - Perpignan
  - Pessac
  - Pointe à Pitre
  - Pontoise
  - Quimper
  - Rennes
  - Rouen
  - Saint-Denis
  - Saint-Dizier
  - Saint-Pierre
  - Strasbourg
  - Suresnes
  - Toulon
  - Toulouse
  - Tours
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Villejuif